CLINICAL TRIAL: NCT03665766
Title: The Effect of Cyclosporine A Versus Tacrolimus on the Response to Antiviral Treatment After HCV Genotype -4 Recurrence in Recipients of Living Donor Liver Transplantation
Brief Title: Effect of Cyclosporine A Versus Tacrolimus on Response to Antiviral Therapy After Hepatitis C Genotype -4 Recurrence Post Liver Transplantation
Status: Completed | Type: Observational
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Iman Fawzy Montasser, Associate professor -Tropical medicine-faculty of medicine-Ain Shams University, Ain Shams University
Other Study IDs: ASU-1124568
Record Dates: First submitted 2018-09-07; First posted 2018-09-11 (Actual); Last update posted 2018-09-11 (Actual); Status verified 2018-09

CONDITIONS: Liver Transplantation
MeSH Terms: interventions — Cycloserine; Tacrolimus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: Yes

GROUPS / COHORTS (6):
- IFN group received Cyclosporine: Living donor liver transplantation recipients with recurrent HCV received Peg IFN-α 2a and RBV as antiviral therapy and Cyclosporine A as primary immunosuppression ,this was routinely taken not as intervention according to local practice
  Interventions: Drug: Cycloserine,Tacrolimus
- IFN group received tacrolimus: Living donor liver transplantation recipients with recurrent HCV received Peg IFN-α 2a and RBV as antiviral therapy and Tacrolimus as primary immunosuppression ,this was routinely taken not as interventing according to local practice
  Interventions: Drug: Cycloserine,Tacrolimus
- Sof plus Rbv group received Cyclosporine: Living donor liver transplantation recipients with recurrent HCV received sofosbuvir and RBV as antiviral therapy and Cyclosporine as primary immunosuppression,this was routinely taken not as intervention according to local practice
  Interventions: Drug: Cycloserine,Tacrolimus
- Sof plus Rbv received tacrolimus: Living donor liver transplantation recipients with recurrent HCV received sofosbuvir and RBV as antiviral therapy and Tacrolimus as primary immunosuppression,this was routinely taken not as intervention according to local practice
  Interventions: Drug: Cycloserine,Tacrolimus
- Sof,dac pus ribavirin received cyclosporine: Living donor liver transplantation recipients with recurrent HCV received daclatasvir, sofosbuvir and RBV as antiviral therapy and Cyclosporine as primary immunosuppression,this was routinely taken not as intervention according to local practice
  Interventions: Drug: Cycloserine,Tacrolimus
- sof,dac plus rbv received tacrolimus: Living donor liver transplantation recipients with recurrent HCV received daclatasvir, sofosbuvir and RBV as antiviral therapy and Tacrolimus as primary immunosuppression,this was routinely taken not as intervention according to local practice
  Interventions: Drug: Cycloserine,Tacrolimus

INTERVENTIONS:
Drug: Cycloserine,Tacrolimus

SUMMARY:
Background and Aim: The immunosuppression influence on the response to antiviral therapy (AVT) for recurrent hepatitis C virus (HCV) infection in liver transplant (LT) recipients remains controversial, especially for the rarely investigated genotype 4.This study aims to compare the effects of the two widely used calcineurin inhibitors(CNIs)(Cyclosporine A (CsA) and tacrolimus (Tac)) on the therapeutic response to different AVT regimens. Method: In126 living donor liver transplant (LDLT) recipients with recurrent HCV infection, participants were categorized to three groups according to AVT. Group one received pegylated interferon (Peg IFN-α 2a) and ribavirin (RBV) (n= 44), group two received the direct antiviral agent (DAA) sofosbuvir plus RBV (n=52) and group three received daclatasvir, sofosbuvir (other DAAs) plus RBV(n=30) each group was further subdivided according to primary immunosuppression (CsA or Tac). The sustained virological response (SVR) and relapse rates were considered the primary therapeutic outcomes of AVT. The virological response guided therapy end points for AVT were considered the secondary outcomes.

ELIGIBILITY:
Inclusion Criteria:group(I):participants received Peg IFN-α 2a and RBV therapy who fulfilled the following inclusion criteria:

* Age between 18 and 65 years ;
* elevated aminotransferase levels (ALT and AST)
* detectable HCV RNA by polymerase chain reaction (PCR)
* liver biopsy results consistent with HCV recurrence using the Metavir scoring system (Metavir ≥A1F1)
* For group II and III:
* age between 18 and 75 years
* detectable HCV RNA by PCR

Exclusion Criteria:group I

* if they were younger than 18 years or older than 65 years or had one of the following criteria
* alcoholic
* poorly controlled autoimmune disease
* significant cardiac disease
* suicidal ideation
* a history of suicide attempt
* major psychosis
* serum creatinine ˃3 mg/dl
* thyroid dysfunction
* combined kidney-liver transplantation
* were currently pregnant or planning pregnancy.

Group II and III:

* younger than 18 years or older than 75 years
* total bilirubin (T.Bil) >3 mg/dl
* serum albumin< 2.8 mg/dl
* international normalized ratio ≥1.7
* Platelet count < 5000/mm3
* HCC, except 4 weeks after intervention with no evidence of activity using computed tomography or magnetic resonance imaging
* extra hepatic malignancy except after two years of disease free-interval
* uncontrolled diabetes evidenced by glycated haemoglobin >9%
* were pregnant .

Ages: 18 Years to 75 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: living donor liver transplant (LDLT) recipients with recurrent HCV infection, participants were categorized to three groups according to AVT. Group one received pegylated interferon (Peg IFN-α 2a) and ribavirin (RBV) , group two received the direct antiviral agent (DAA) sofosbuvir plus RBV and group three received daclatasvir, sofosbuvir (other DAAs) plus RBV each group was further subdivided according to primary immunosuppression (CsA or Tac)
Sampling Method: Non-Probability Sample
Enrollment: 126 (Actual)
Dates: Start 2014-05-15 (Actual); Primary Completion 2018-04-02 (Actual); Study Completion 2018-04-02 (Actual)

PRIMARY OUTCOMES:
sustained virological response | 24 weeks for group I and 12 weeks for group II and III
  a negative serum HCV RNA